CLINICAL TRIAL: NCT06812091
Title: Prediction and Treatment of Pediatric Diseases and Long-term Outcomes Through Microbiome and Multi-Omics Study by Life Cycle
Brief Title: Human Microbiome Research and Development for Overcoming Pediatric Diseases
Status: Recruiting | Type: Observational
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Hyun-Kyung Park, Professor, MD, PhD, Hanyang University
Other Study IDs: HYUMC IRB No. 2023-04-047
Record Dates: First submitted 2025-01-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Human Microbiome; Pediatrics; Disease; Growth & Development
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — fecal DNA extraction and storage for NGS analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prediction and treatment of pediatric diseases and long-term outcomes through microbiome and multi-omics analysis by life cycle: We aim to demonstrate that a wide range of diseases are associated with gut microbiome dysbiosis and to investigate the subsequent recovery (restoration) or further deterioration of the gut microbiome over time. This study seeks to offer a novel perspective on changes in the gut microbiome, particularly in the context of the gut-lung and gut-brain axes.

DETAILED DESCRIPTION:
Fecal samples are collected and analyzed from birth through childhood, including those from both preterm and term infants. Based on these collected samples, groups are categorized into disease groups commonly observed in children. Genomic DNA is extracted from the fecal samples, followed by high-throughput 16S rRNA amplicon sequencing to analyze the microbial composition. Additionally, multiomics analyses, including metabolomics, are conducted to provide a comprehensive understanding of gut microbiome dynamics. The impact on the microbiome is further investigated in vitro using a fermenter-based intestinal microbiota model system.

ELIGIBILITY:
Inclusion Criteria:

* children (including newborns) who have obtained their consent from their guardians

Exclusion Criteria:

* subjects who did not obtain consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Control group: healthy infants without any diagnosed diseases, born full-term, exhibiting normal growth and development.
  Case group: infants with diagnosed diseases, including those born prematurely, those with a history of neonatal intensive care unit (NICU) admission, and those exhibiting neurodevelopmental impairments.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Follow-up of growth percentile in height, weight, and head circumference | 2 months old, 4 months old, 6 months old, 1 year old, and then every year until the age of ten years
  Monitoring the baby's growth status compared to the Nomogram growth chart
Obervation of age-specific developmental milestones | 4 months old, 1 year old, 3 years old, school age
  Judging whether the development status is appropriate according to developmental milestones based on developmental screening tests and doctors' opinions)
Observations on the incidence and frequency of enteritis, sepsis, and respiratory diseases | 2 months old, 4 months old, 6 months old, 1 year old, and then every year until the age of ten years
  The dysbiosis of the gut microbiome affects various organs, such as the gut-lung axis and the gut-brain axis, in addition to the disease of the intestine itself, so monitor the occurrence of infectious diseases

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Kyung Park, MD, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea